CLINICAL TRIAL: NCT05139043
Title: Safety and Imaging of Post-Operative Low Dose Versus Standard Dose Dexamethasone in Patients with Primary or Metastatic Brain Tumors: a Randomized, Double-blinded Feasibility Study.
Brief Title: Low Dose Versus Standard Dose Dexamethasone for Reduction of Swelling in Patients with Primary or Metastatic Brain Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20624; NCI-2021-11292 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20624 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2021-12-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Malignant Brain Neoplasm; Metastatic Malignant Neoplasm in the Brain; Recurrent Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard dose dexamethasone) (Active Comparator): Patients receive standard dose dexamethasone PO q 12 h for 3 days. On the day of surgery, patients receive standard dose dexamethasone IV before and after the surgery. Patients receive standard dose dexamethasone IV q 12 h on days 1-3 post surgery and tapered dexamethasone PO q 12 h on days 4-14 in the absence of disease progression or unacceptable toxicity. Additional doses of dexamethasone are given if needed.
  Interventions: Drug: Dexamethasone
- Arm II (lower dose dexamethasone) (Experimental): Patients receive lower dose dexamethasone PO q 12 h for 3 days. On the day of surgery, patients receive lower dose dexamethasone IV before and after the surgery. Patients receive lower dose dexamethasone IV q 12 h on days 1-3 post surgery and tapered dexamethasone PO q 12 h on days 4-14 in the absence of disease progression or unacceptable toxicity. Additional doses of dexamethasone are given if needed.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Given IV and PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex

SUMMARY:
This phase II trial studies whether low dose dexamethasone works as well as standard dose dexamethasone to reduce brain swelling after brain surgery in patients with primary brain tumors or cancer that has spread from other places in the body to the brain (metastatic). Surgery is an important part of the treatment of brain tumors; however, it results in injury to surrounding brain tissue, leading to brain swelling. Dexamethasone is effective for controlling the swelling of the brain; however, dexamethasone can cause many unwanted side effects. To minimize the side effects of dexamethasone, the lowest dose needed to control swelling of the brain should be used. This research study is assessing the safety of using a lower than standard dose of dexamethasone after the surgery to control brain swelling.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of administering lower doses of dexamethasone post-operatively in patients who have mild to moderate cerebral edema pre-operatively.

II. Describe the toxicity profile associated with post-operative lower doses and standard doses of dexamethasone, separately.

SECONDARY OBJECTIVES:

I. Descriptively assess the consistency between the quantitative data produced by strategically acquired gradient echo (STAGE) and qualitative assessments of changes in cerebral edema on serial fluid-attenuated inversion recovery (FLAIR) images.

II. Quantitatively assess changes in the volume of cerebral edema post-operatively in participants on Arm 1 (standard dose) and Arm 2 (low dose).

EXPLORATORY OBJECTIVE:

I. Describe changes in the volume of cerebral edema between pre-operative and post-operative day 1 brain magnetic resonance imaging (MRIs) in Arm 1 (standard dose) and Arm 2 (low dose) participants, separately.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard dose dexamethasone orally (PO) every 12 hours (q 12 h) for 3 days. On the day of surgery, patients receive standard dose dexamethasone intravenously (IV) before and after the surgery. Patients receive standard dose dexamethasone IV q 12 h on days 1-3 post surgery and tapered dexamethasone PO q 12 h on days 4-14 in the absence of disease progression or unacceptable toxicity. Additional doses of dexamethasone are given if needed.

ARM II: Patients receive lower dose dexamethasone PO q 12 h for 3 days. On the day of surgery, patients receive lower dose dexamethasone IV before and after the surgery. Patients receive lower dose dexamethasone IV q 12 h on days 1-3 post surgery and tapered dexamethasone PO q 12 h on days 4-14 in the absence of disease progression or unacceptable toxicity. Additional doses of dexamethasone are given if needed.

After completion of surgery, patients are followed up after 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years or older.
* Participant has a Karnofsky Performance Status of >= 60%.
* Participant has a primary or metastatic brain tumor(s).
* Participant can have newly diagnosed or recurrent brain tumor(s).
* If a participant is requiring more than 3 mg orally every 12 hours (q 12 h) of dexamethasone at the time of signing the consent form, it is anticipated by the neurosurgeon that the participant will be able to taper down their dose of dexamethasone to 3 mg orally q 12 h by 3 days before the surgery.

  * (Note: If the patient is not able to decrease their dose of dexamethasone to 3 mg orally q 12 h 3 days before surgery, the patient will not be allowed to participate in the study.)
* Participant must have less than 10 mm of midline shift seen on pre-op brain magnetic resonance imaging (MRI).
* The neurosurgeon anticipates being able to perform a gross total resection of tumor.
* Participant is not planning to participate in another clinical trial during the study period.
* There is no limit to the number of prior therapies for enrollment in this study.
* All participants must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Participant is unable to undergo a brain MRI.
* Participant is unable to tolerate dexamethasone.
* Participant has a chronic or active viral infection of the central nervous system (CNS).
* Participant has a coagulopathy or bleeding disorder.
* Participant has an uncontrolled illness including ongoing or active infection.
* Participant has another active malignancy.
* A patient has a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the safety monitoring requirements and completion of treatment according to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-09 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Lack of feasibility | Up to post-operative day 8
  Defined as a participant requiring more than 18 mg of dexamethasone beyond the planned dose per treatment arm during the 9 day period from surgery through post-operative day 8. Feasibility will be monitored sequentially (after each patient completes study treatment), by arm. The feasibility review boundary is based on a Wald sequential probability ratio test. Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Incidence of toxicity | Up to 30 days
  All grade toxicities attributed to dexamethasone at the possible or above level. All toxicities and side effects will be summarized in tables by organ, severity, and attribution. Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.

SECONDARY OUTCOMES:
Volume of cerebral edema for each post-surgery brain magnetic resonance imaging (MRI) | Up to 30 days
  Measured by strategically acquired gradient echo (STAGE).
Qualitative assessments of cerebral edema on serial fluid-attenuated inversion recovery (FLAIR) images for each post-surgery brain MRI | Up to 30 days
  Descriptive statistics will be provided for cerebral edema volume as measure by STAGE for each arm by strata and time point.

OTHER OUTCOMES:
Volume of cerebral edema for pre-operative and post-operative day 1 brain MRIs as measured by STAGE | At pre-operative and post-operative day 1
  Descriptive statistics will be provided for cerebral edema volume as measure by STAGE for each arm by strata and time point.
Qualitative assessments of cerebral edema on serial FLAIR images for pre-operative and post-operative day 1 brain MRIs | At pre-operative and post-operative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jana L Portnow, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States